CLINICAL TRIAL: NCT01310673
Title: Therapy for Acute Gout: Does Initial Use of Allopurinol Effect Duration and/or Recurrence Rate of Acute Attacks
Brief Title: Initiation of Allopurinol at First Medical Contact for Acute Attacks of Gout
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Thomas H. Taylor MD, Chief Rheumatology and Infectious Diseases, White River Junction VA Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPHS #16820
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Gout; Gout Acute
Keywords: Gout; Allopurinol; Acute gout
MeSH Terms: conditions — Gout | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allopurinol (Active Comparator)
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Allopurinol — Allopurinol 300mg po QD for 30 days.
  Indomethacin 50mg TID for 10 days. Colchicine 0.6mg po Bid or QD, as tolerated for 90 days.
  Arms: Allopurinol
Drug: Placebo — Placebo tablet QD for 10 days, followed by delayed allopurinol 300mg po QD days 11-30.
  Indomethacin 50mg TID for 10 days. Colchicine 0.6mg po Bid or QD, as tolerated for 90 days.
  Arms: Placebo

SUMMARY:
Medical teaching suggests allopurinol should not be initiated in the setting of an acute attack of gout, as rapid lowering of serum urate may exacerbate the attack. This study tests the hypothesis that there is no difference in patient reported daily pain or flair occurrences with early versus delayed institution of allopurinol during an acute gout attack.

DETAILED DESCRIPTION:
Design: Randomized, placebo-controlled, double-blind trial. Setting: Outpatient clinics, White River Junction Veterans Affairs Medical Center.

Patients: 57 men with crystal proven acute gout attack, at first medical contact, and within 7 days onset.

Intervention: Subjects were randomized to receive allopurinol 300mg daily or matching placebo for 10 days. All patients received indomethacin 50mg TID for 10 days, prophylactic dose colchicine 0.6mg BID for 90 days, and open-label allopurinol starting at day 11.

Measurements: Primary outcomes were patient reported pain on visual analogue scale (VAS) for the primary joint, and self reported flares in any joint days 1-30. Secondary endpoints included urate, sedimentation rates, C-reactive protein levels.

ELIGIBILITY:
Inclusion Criteria:

* First medical contact for acute attack of gout.
* ACR criteria for acute attack of gout
* Crystal proven by arthrocentesis on day of enrollment
* Primary gout

Exclusion Criteria:

* Secondary Gout
* Tophaceous Gout
* Prior steroid, colchicine, or uric acid lowering therapy in the past 6 months.
* Uncontrolled CHF
* Unstable angina
* Renal insufficiency (entry CREAT > 1.3)
* Anticoagulant therapy
* Immunosuppressive therapy or chemotherapy in the past 6 months
* Pregnancy; OR
* Known allergy to NSAID, colchicine, or allopurinol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 1998-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Daily pain scores and recurrence attack rate. | 30 days after initiation of treatment
  Daily pain measured on a visual analogue scale over 10 days after initiation of treatment.
  Patient reported gout recurrences over 30 days

SECONDARY OUTCOMES:
sedimentation rates and C-reactive protein at 0, 3, 10, and 30 day visits | 30 days
  Fall in ESR and CRP were measured as confirmation of attack resolution

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Taylor, MD, Principal Investigator — White River Junction VA Medical Center
Locations (1):
- White River Junction VA Medical Center, White River Junction, Vermont, United States

REFERENCES:
- [Derived] Taylor TH, Mecchella JN, Larson RJ, Kerin KD, Mackenzie TA. Initiation of allopurinol at first medical contact for acute attacks of gout: a randomized clinical trial. Am J Med. 2012 Nov;125(11):1126-1134.e7. doi: 10.1016/j.amjmed.2012.05.025. PMID 23098865